CLINICAL TRIAL: NCT01850576
Title: Project Tailoring Effective And Community-based HIV Interventions in Kenya
Brief Title: Project TEACH-Kenya
Acronym: TEACH
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We did not receive proper funding to complete this study
Sponsor: North Bronx Healthcare Network (Other)
Responsible Party: Principal Investigator, Yvette Calderon,MD, MS, Principal Investigator, North Bronx Healthcare Network
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2013-PA-12-231
Record Dates: First submitted 2013-05-02; First posted 2013-05-09 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: HIV
Keywords: prevention; testing; counseling; linkage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Those randomized to the intervention group will be invited to attend the risk reduction intervention.
  Interventions: Behavioral: Risk Reduction Intervention
- Control (No Intervention): The control group will receive usual care. Both treatment and control groups will have received the video-based risk reduction intervention.

INTERVENTIONS:
Behavioral: Risk Reduction Intervention — STEP is based on social learning theory and provides age-appropriate and culturally acceptable HIV prevention information in a format that encourages information growth and skills enhancement. The program is delivered by 'Instructors,' undergraduate college students aged 18-24, one hour per week for 10 weeks.
  Arms: Intervention

SUMMARY:
Public health programs and policies have utilized the "combination prevention" model of bringing together tailored, proven interventions in order to reduce the global impact of HIV. Project TEACH-Kenya adapts two effective HIV interventions, Project BRIEF (Behavioral intervention, Rapid HIV test, Innovative video, Efficient cost and health care savings, Facilitated seamless care) and STEP (Skill-based Teenage Education Program for HIV prevention) to increase HIV testing and counseling rates, implement proven risk reduction programs, and improve rates of linkage to care and ART initiation among adolescents in Kenya. The collaboration with St. Francis Community Hospital and input from the Kasarani community will increase the breadth, reach, and impact of this HIV prevention intervention in Kenya.

DETAILED DESCRIPTION:
In 2010, HIV/AIDS accounted for up to 29% of all deaths and 24% of all disabilities in Kenya. There is a particular need to concentrate HIV education, testing, and linkage-to-care efforts among high-risk adolescents; by age 18, 47% of women and 58% of men have had sexual intercourse. Only one in four young Kenyans used condoms the first time they had sex, and only half of 15-24 year olds had comprehensive HIV knowledge. The goal of this intervention, Project TEACH-Kenya, is to adapt two proven HIV interventions, Project BRIEF and STEP, to an urban setting in the Kasarani District of the Nairobi Province, Kenya. According to the US President's Emergency Plan for AIDS Relief (PEPFAR) Five-Year Strategy, a successful prevention program brings together a combination of evaluated, tailored interventions, to stem the spread of HIV infection among high-risk populations. This synergistic model, referred to as combination prevention, serves as the basis for adapting the current intervention encompassing HIV testing and counseling, risk behavior reduction programs, and linkage to care and ART initiation to the Kenyan context. Project TEACH-Kenya will develop tailored, theory-based educational videos, linkage procedures, and a tailored prevention program for adolescents 13-18 years old and pilot and test the intervention at St. Francis Community Hospital, a high volume community-based hospital in Kasarani. The majority of adolescents that access St. Francis's services are orphan and vulnerable children affected by HIV/AIDS (OVC-HIV) who are disproportionately poor and malnourished and are at increased risk for acquiring HIV, stressing the need for this intervention. The outcome of this project will be a feasible, evidence-based, cost- and time-effective program to improve HIV education and increase testing and linkage-to-care rates among adolescents in Kenya.

ELIGIBILITY:
Inclusion Criteria:

* Women and minorities will not be excluded from this research study. We will include only adolescents ages 13-18 at time of recruitment in this study, because that is the age group that we are targetting for this intervention. Residents must be of the St. Francis Hospital catchment area

Exclusion Criteria:

* Over the age of 18 and under the age of 13. Unable to understand the consent process for the study; or otherwise unable to consent to HIV testing.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2013-09; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Feasibility | up to 15 months
  Feasibility of implementing project STEP will be measured by acceptance and participation rates. Evaluation outputs include:
  1. Efficiency: Number of eligible participants, number randomized into each age and experimental group,
  2. Acceptance rates (number of people who agree to participate in program; number who complete the whole 10 week program);
  3. Population characteristics: We will describe the demographic and behavioural profiles of those who participated in the program and those who refuse; the level of HIV knowledge, self efficacy and satisfaction with the program.
  4. Satisfaction/acceptability: College student recruitment, receptivity and satisfaction with the project; implementation issues and resource use

SECONDARY OUTCOMES:
Risk Reduction | up to 15 months
  HIV related knowledge will be measured using the HIV KQ-18; stigma will be measured using the AIDS-Related Stigma Scale. Sexual history will also be measured using the traditional Project B.R.I.E.F. survey. The questionnaire will be piloted for receptiveness. We will ask for ratings of satisfaction with the video-based pre-counseling and education/prevention post test using measures used by Calderon.

CONTACTS AND LOCATIONS:
Overall Officials: Rosy Chhabra, PsyD, Principal Investigator — Albert Einstein College of Medicine; Yvette Calderon, MD, MS, Principal Investigator — North Central Bronx Healthcare Network; Erick Nyambedha, Study Director — St. Francis Community Hospital
Locations (2):
- Albert Einstein College of Medicine, The Bronx, New York, United States
- St. Francis Community Hospital, Nairobi, Kasarani, Kenya